CLINICAL TRIAL: NCT05513508
Title: A Pragmatic Open Label, Multi-center, Spontaneous, No-profit, Randomized Controlled Clinical Trial With Non-significant Risk Medical Device on the Rotational Use of Interfaces Versus Standard of Care for Patients Treated With NPPV for AHRF.
Brief Title: The ROTAtional-USE of Interface STUDY
Acronym: ROTA-USE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Collaborators: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Principal Investigator, Rosanna Vaschetto, MD, PhD, Associate Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 062.373
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Pressure Ulcer; Noninvasive Positive Pressure Ventilation; Acute Hypercapnic Respiratory Failure
Keywords: Rotational use of noninvasive interfaces
MeSH Terms: conditions — Pressure Ulcer; Respiratory Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the intervention group the first mask will be randomly chosen between the two most used in that center among those available i.e., oro-nasal, total face or hybrid mask. Thereafter, NPPV mask will be changed every 6 hours, alternating the two different interfaces. Patients wearing oro-nasal masks will receive protective dressings on nasal bridge before starting NPPV.
  Interventions: Procedure: Protocolized rotational use of interfaces
- Control group (Active Comparator): In the control group, mask will be chosen according to the standard of care of the participating centers among the three types of masks available i.e., oro-nasal, total face or hybrid mask. Patients wearing oro-nasal masks will receive protective dressings on nasal bridge before starting NPPV. Interface will be changed in case of discomfort judged by the patient as unbearable or in case of the presence of a pressure sore.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Procedure: Protocolized rotational use of interfaces — The NIV mask will be changed every 6 hours, alternating two different interfaces between the two most used in that center among those available i.e., oro-nasal, total face or hybrid mask.
  Arms: Intervention group
Procedure: Standard of care — Mask will be chosen according to the standard of care of the participating centers among the three types of masks available i.e., oro-nasal, total face or hybrid mask. Interface will be changed in case of discomfort judged by the patient as unbearable or in case of the presence of a pressure sore.
  Arms: Control group

SUMMARY:
In this trial investigators will explore if a protocolized rotational use of interfaces i.e., masks, during noninvasive positive pressure ventilation (NPPV) compared to standard care is clinically effective and cost-effective in reducing the incidence of pressure sores in patients with hypercapnic acute respiratory failure (AHRF) treated continuously i.e., for more than 24 hours, with NPPV (to avoid intubation, as alternative to invasive ventilation and after early extubation and weaning).

DETAILED DESCRIPTION:
Objectives:

Primary objective To determine if a protocolized rotational use of interfaces during NPPV compared to standard care is effective in reducing the development of new pressure sores in patients with hypercapnic ARF treated continuously i.e., for more than 24 hours, with NPPV (to avoid intubation, as alternative to invasive ventilation, and during early extubation and weaning).

Measurements of effectiveness include:

The primary effectiveness outcome will be the proportion of patients who develop new pressure sores at 36 hours from randomization. Secondary outcomes will be the onset of pressure sores measured at different time points (12, 24, 36, 48, 60, 72, 84, 96 hours), number and stage of pressure sores and comfort measured at the same time points of the primary outcome. The location of pressure sores per patient will be also collected. The study will also monitor the number of patients that will interrupt NPPV treatment for discomfort, the presence of eyes irritation, the adherence to the protocol (duration of NPPV treatment/day, interface change, hygiene protocol application) and the presence of vasoactive medications. Variables like nutritional status at randomization, Braden Scale and Frailty Index at hospital entrance, total duration of NPPV from randomization, duration of NPPV per day, hospital length of stay and in-hospital mortality will be recorded. The economic impact of the protocolized rotational use of interfaces will be assessed through a cost-effectiveness analysis evaluating the additional costs needed to avoid a pressure sore due to the planned intervention as well as the costs needed to actively treat skin ulcers due to failure of preventing measures in both groups of patients.

Randomization:

A 1:1 stratified randomization will be performed to assigned patients to the protocolized rotational use of interfaces (experimental treatment) or standard of care (comparison group). Subjects will be stratified according to center and ward (intensive care unit, intermediate respiratory care unit, respiratory medicine service or internal medicine service according to hospital organization). Within each stratum, subjects will be randomly assigned to one of the treatments using a predefined randomization list. To ensure masking, randomization schemes will be input directly into the Research Electronic Data Capture (REDCap) system. In the treatment group, the first interface will be randomly assigned. Randomization scheme will be input directly into REDCap system.

Study treatments:

In both arms, the treatment according to the assigned protocol will be continued until patients require NPPV.

Skin underneath the mask and occipital region, will be inspected every 12 hours to check for any possible damage by assessors blind to the study protocol. Assessors (physicians or nurses) will be instructed to recognize pressure sores and their stage. Before starting the study recruitment, the assessors will take a test aiming to correctly stage 10 pressure sores. Only assessors who will recognize all of them, participate to the study. Test will be taken trough google forms and results will be registered for the study. To minimize detection bias, assessors will not participate to the care of the patient and will be blind on patient group of assignment. If a pressure sore will be detected, physician in charge of the patient will be promptly informed and a note will be written on the nursing record.

Pressure sores will be stage as follows:

stage I: A reddened, painful area on the skin that does not turn white when pressed. This is a sign that a pressure ulcer may be forming. The skin may be warm or cool, firm or soft.

stage II: The skin blisters or forms an open sore. The area around the sore may be red and irritated.

stage III: The skin now develops an open, sunken hole called a crater. The tissue below the skin is damaged. You may be able to see body fat in the crater.

stage IV: The pressure ulcer has become so deep that there is damage to the muscle and bone, and sometimes to tendons and joints.

In addition to the 4 main stages for pressure sores, there are 2 others: 1) "Unstageable" is when you can't see the bottom of the sore, so you don't know how deep it is; 2) "Suspected Deep Tissue Injury" when the surface of the skin looks like a Stage 1 or 2 sore, but underneath the surface it's a Stage III or IV.

Discomfort due to the mask will be evaluated every 12 hours using a 5-level Likert-like scale to answer the questions "How is your level of discomfort related to the mask?" (in Italian). The extremes of the scale are "1 - no discomfort" and "5 - unbearable discomfort," with three intermediate levels ("light discomfort," "moderate discomfort," and "intense discomfort").

NPPV standard management:

In both arms, standard care (diagnostic tests, administration of systemic therapy including antibiotics, steroids and inhaled bronchodilator therapy and hemodynamic management) will be applied according to the clinical practice of each institution.

The right size of the mask will be selected according to the indications provided by the manufacturer. The mask straps will be adjusted according to the " two-finger rule " not to tighten to hard the headgear.

Following international guidelines, patients who benefit from NPPV during the first four hours of treatment will receive NPPV for as long as possible during the first 24 hours. Target saturation range will be 88-92% either spontaneously breathing or when receiving NPPV. NPPV treatment will last until the acute cause has resolved, commonly about two to three days.

NPPV will be started as suggested by the British Thoracic Society/Intensive Care Society Guideline for the ventilatory management of AHRF in adults. NIV will be started when pH <7.35 and PaCO2 >6.5 kilopascal (kPa) persist or develop despite optimal medical therapy, targeting an oxygen saturation of 88-92%. Blood gas exchange will be performed before starting NPPV treatment and after 2 hours from its starting and thereafter, when clinically indicated. NPPV will be initially set in a pressure support mode with a ventilator designed specifically to deliver NPPV or with an ICU ventilator provided with noninvasive ventilation mode. Expiratory positive airway pressure (EPAP) will be set at 3-5 Centimeters of Water (cmH2O) while inspiratory positive airway pressure (IPAP) will be set to achieve adequate augmentation of chest/abdomen movement with an expiratory tidal volume of 6-8ml/kg and a reduction of respiratory rate (< 30 breath/min) together with a good patient ventilator interaction (i.e., pressure-flow curve monitoring). The presence of active humidification will be left to the choice of the doctor in charge for that patient, although heated humidification should be considered if the patient complains of mucosal dryness or if respiratory secretions are thick and tenacious.

The weaning strategy will be documented in the medical and nursing records. The following might be use as general indication: continue NPPV for 16 hours on day 2; 12 hours on day 3 including 6-8 hours overnight use; NPPV may be discontinued on day 4 unless continuation is clinically indicated.

The suggested monitoring during NPPV will be continuous peripheral oxygen saturation, intermittent measurement of PaCO2 and pH, ECG monitoring in the patient with a pulse rate >120 bpm or if there is dysrhythmia or possible cardiomyopathy.

As guidelines recommend keeping the skin dry and clean under medical equipment, a protocol for skin will be adopted by all centers included in the study.

If a patient needs prolonged continuous NPPV, brakes will be programmed and annotated in the case report form, in case of instability, interface will be removed for about 10 minutes only to ensure oxygenation.

When signs of skin trauma become apparent, a barrier dressing and a strategy of regular breaks and alternating between two interface types will be used. In case of mask-related rash even in the absence of allergy, topical steroids may be indicated and/or antibiotics if the wound becomes infected. In case NPPV causes severe gastric distension, a nasogastric tube will be inserted.

Early extubation and weaning with NPPV:

According to the guidelines, NPPV is recommended to aid weaning from invasive mechanical ventilation in patients with AHRF, secondary to COPD and to other causes of AHRF, when local expertise in its use exists. Patients during invasive mechanical ventilation will be treated according to the clinical guidelines. After setting maximum medical treatment, once with ventilation in a controlled mode pH and PaCO2 will be normalized in presence of neurological, hemodynamic and respiratory stability, patients will be extubated and put in NPPV. The ventilator will be set with the same positive end expiratory pressure (PEEP) and inspiratory pressure support (PS) level applied during invasive mechanical ventilation, setting the fastest pressure rise time at least during the first 24 hours after extubation. Then, NPPV will be gradually withdrawn if patients tolerated spontaneous breathing until they could permanently sustain spontaneous breathing.

Data collection:

A RedCap database will be set up to collect the information needed for the study. The database will be made of 10 sheets: the first one collecting the baseline demographic and clinical characteristics of the patients and the others will be made to collect the outcomes' information at each time point and a discharge sheet including information on the overall treatment.

The randomization procedure will be implemented within Redcap.

Sample size:

Given a type I error of 0.05, a power of 0.8, an expected proportion of patients who develop pressure sores in the control group of 23% and an expected dropout rate of 5%, 239 subjects per group are estimated to identify a 10% absolute difference in the proportion of patients developing pressure sores between intervention and control groups measured at 36 h from randomization.

Statistical analysis:

The analyses will be performed according to the intention to treat principle. Descriptive statistics will be calculated to summarized patient characteristics collected at study entry according to randomization group. Categorical variables will be reported as absolute frequencies and percentages and continuous variables as mean and standard deviation or median first and third quartiles if not normally distributed according to the Shapiro-Wilks test.

The raw risk of pressure sore will be calculated ad each time point as the ratio between the number of subjects who developed a pressure sore at the time point divided by the number of subjects undergoing NPPV at the time point. Patients having a planned break at the time-point considered, but not been weaned off the NPPV treatment yet, will be considered undergoing NPPV.

Mixed effect logistic regression models will be used to estimate the risk of pressure sores and the difference between interfaces including a random intercept to account for clustering of the subjects within center and repeated measures within patients. The response variable will be the presence/absence of pressure sores and the independent variables the treatment, time (12, 24, 36, 48, 60, 72, 84, 96) and their interaction. The marginal and center specific predicted probabilities estimated by the model will provide the incidence of pressure sores at different times and overall. The inclusion of time as covariate will allow to test the presence of a time trend in incidence of pressure sores and to investigate the variation of time trends according to treatment group.

Regarding the number of pressure sores, different mixed effect Poisson regression models will be applied: one for each time point to estimate the average number of pressure sores at each time point and a model in which only the highest number of pressure sores will be considered for each patient. Time will be included as offset to evaluate the average number of pressure sores per day.

The grade and location of pressure sores will be summarize using descriptive statistics at each time point.

Regarding the economic evaluation. the incremental cost effectiveness ratio (ICER) will be calculated considering two outcomes: i) the proportion of pressure sores and ii) the comfort. The ICER as the ratio between the difference each outcome in the two groups (difference in the proportion of pressure sores or comfort score) and the difference in the average cost for each treatment allowing to evaluate the incremental costs needed to reduce of 1 point the outcomes thanks to the rotational use of interfaces. The confidence intervals of the ICER will be calculated using the non-parametric bootstrap method, specifically the 2.5th and 9.75th percentiles of the bootstrap distribution of ICER will be considered as the lower and higher limits of the confidence interval. The cost-effectiveness acceptability curve will be also drawn to evaluate the probability of the intervention to be cost-effective considering different thresholds.

Safety monitoring:

A single interim analysis will be performed when a number of patients equal to two-thirds of the predefined sample are randomized and complete the study. Early stopping criteria will be a predetermined 2-sided p value < 0.01 for the rejection of the null hypothesis that the strategies are equivalent in terms of rate of pressure sores.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Patients with chronic obstructive pulmonary disease (COPD) exacerbation or with AHRF of a different etiology needing NPPV to avoid intubation (pH < 7.35 with PaCO2 > 45 mmHg and partial pressure of oxygen (PaO2) < 65 mmHg plus respiratory rate > 25 breath/min with clinical signs of respiratory muscle distress); or as alternative to invasive ventilation with a forecast of treatment of at least 24 hours admitted to the intensive care unit, intermediate respiratory care unit, respiratory medicine service or internal medicine service according to hospital organization; or patients with chronic pulmonary disease intubated for a COPD exacerbation or for pneumonia who are early extubated and weaned in the intensive care unit with NPPV with a forecast of treatment of at least 24 hours.

Exclusion Criteria:

* Patient with skin breakdown or non-blanchable erythema in one of the following areas i.e., nasal bridge, nasolabial fold, cheek or scalp at hospital entrance;
* Patients who refuse to consent to the study protocol;
* Patient known to be pregnant;
* Patients with contraindication to NPPV (lack of spontaneous breathing; gasping; anatomical or functional airway obstruction; gastrointestinal bleeding or ileus; coma; massive agitation; massive retention of secretions despite bronchoscopy and aggressive physiotherapy; hemodynamic instability (cardiogenic shock, myocardial infarction); status post upper gastrointestinal surgery);
* Patients entering hospital with asthma, with cardiogenic pulmonary edema;
* Patients with tracheostomy;
* Patients needing NPPV only for palliation of symptoms (relief of dyspnea) i.e., category 3 defined by the Task Force on the Palliative Use of NPPV of the Society of Critical Care Medicine;
* Use of high flow nasal cannula integrated with NPPV for weaning strategy;
* Pre-existing skin erythematosus diseases;
* Known hypersensitivity to skin protective devices (i.e., polyurethan films, colloids, foams);
* More than 2 hours of NPPV application before randomization;
* Patients already included in the study protocol at an earlier stage of the hospitalization;
* Refuse to wear NPPV interface due to comfort;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who develop new pressure sores | At 36 hours from randomization
  To determine if a protocolized rotational use of interfaces during NPPV compared to standard care is effective in reducing the development of new pressure sores in patients with AHRF treated continuously i.e., for more than 24 hours, with NIV (to avoid intubation, as alternative to invasive ventilation, and during early extubation and weaning).

SECONDARY OUTCOMES:
Onset of pressure sores at different timepoints | At 12, 24, 36, 48, 60, 72, 84, 96 hours from the randomization
  To determine if a protocolized rotational use of interfaces during NPPV compared to standard care is effective in reducing the development of new pressure sores in patients with AHRF treated continuously i.e., for more than 24 hours, with NPPV (to avoid intubation, as alternative to invasive ventilation, and during early extubation and weaning).
Number, stage and location of pressure sores | At 12, 24, 36, 48, 60, 72, 84, 96 hours from the randomization
  Pressure sores will be counted, staged (Stage I, II, III, IV, Unstageable, Suspected Deep tissue Injury) and localized.
NPPV treatment interruption | At 12, 24, 36, 48, 60, 72, 84, 96 hours from the randomization
  The study will also monitor the number of patients that will interrupt NPPV treatment for discomfort, the presence of eyes irritation, the adherence to the protocol (duration of NPPV treatment/day, interface change, hygiene protocol application).
Cost-effectiveness analysis | At 12, 24, 36, 48, 60, 72, 84, 96 hours from the randomization
  The economic impact of the protocolized rotational use of interfaces will be assessed through a cost-effectiveness analysis evaluating the additional costs needed to avoid a pressure sore due to the planned intervention as well as the costs needed to actively treat skin ulcers due to failure of preventing measures in both groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Vaschetto, Assoc, Study Director — Università degli Studi del Piemonte Orientale Amedeo Avogadro
Locations (1):
- Ospedale Maggiore della Carità, Novara, Italy

REFERENCES:
- [Background] Davidson C, Banham S, Elliott M, Kennedy D, Gelder C, Glossop A, Church C, Creagh-Brown B, Dodd J, Felton T, Foex B, Mansfield L, McDonnell L, Parker R, Patterson C, Sovani M, Thomas L. British Thoracic Society/Intensive Care Society Guideline for the ventilatory management of acute hypercapnic respiratory failure in adults. BMJ Open Respir Res. 2016 Mar 14;3(1):e000133. doi: 10.1136/bmjresp-2016-000133. eCollection 2016. No abstract available. PMID 27026806
- [Background] Burns KE, Meade MO, Premji A, Adhikari NK. Noninvasive ventilation as a weaning strategy for mechanical ventilation in adults with respiratory failure: a Cochrane systematic review. CMAJ. 2014 Feb 18;186(3):E112-22. doi: 10.1503/cmaj.130974. Epub 2013 Dec 9. PMID 24324020
- [Background] Vaschetto R, Pecere A, Perkins GD, Mistry D, Cammarota G, Longhini F, Ferrer M, Pletsch-Assuncao R, Carron M, Moretto F, Qiu H, Della Corte F, Barone-Adesi F, Navalesi P. Effects of early extubation followed by noninvasive ventilation versus standard extubation on the duration of invasive mechanical ventilation in hypoxemic non-hypercapnic patients: a systematic review and individual patient data meta-analysis of randomized controlled trials. Crit Care. 2021 Jun 1;25(1):189. doi: 10.1186/s13054-021-03595-5. PMID 34074314
- [Background] Cabrini L, Esquinas A, Pasin L, Nardelli P, Frati E, Pintaudi M, Matos P, Landoni G, Zangrillo A. An international survey on noninvasive ventilation use for acute respiratory failure in general non-monitored wards. Respir Care. 2015 Apr;60(4):586-92. doi: 10.4187/respcare.03593. Epub 2014 Nov 18. PMID 25406347
- [Background] Vaschetto R, Barone-Adesi F, Racca F, Pissaia C, Maestrone C, Colombo D, Olivieri C, De Vita N, Santangelo E, Scotti L, Castello L, Cena T, Taverna M, Grillenzoni L, Moschella MA, Airoldi G, Borre S, Mojoli F, Della Corte F, Baggiani M, Baino S, Balbo P, Bazzano S, Bonato V, Carbonati S, Crimaldi F, Daffara V, De Col L, Maestrone M, Malerba M, Moroni F, Perucca R, Pirisi M, Rondi V, Rosalba D, Vanni L, Vigone F, Navalesi P, Cammarota G. Outcomes of COVID-19 patients treated with continuous positive airway pressure outside the intensive care unit. ERJ Open Res. 2021 Jan 25;7(1):00541-2020. doi: 10.1183/23120541.00541-2020. eCollection 2021 Jan. PMID 33527074
- [Background] Nava S, Navalesi P, Conti G. Time of non-invasive ventilation. Intensive Care Med. 2006 Mar;32(3):361-70. doi: 10.1007/s00134-005-0050-0. Epub 2006 Feb 14. PMID 16477416
- [Background] Mehta S, Hill NS. Noninvasive ventilation. Am J Respir Crit Care Med. 2001 Feb;163(2):540-77. doi: 10.1164/ajrccm.163.2.9906116. No abstract available. PMID 11179136
- [Background] Hess DR. Noninvasive positive-pressure ventilation and ventilator-associated pneumonia. Respir Care. 2005 Jul;50(7):924-9; discussion 929-31. PMID 15972113
- [Background] Tomii K, Seo R, Tachikawa R, Harada Y, Murase K, Kaji R, Takeshima Y, Hayashi M, Nishimura T, Ishihara K. Impact of noninvasive ventilation (NIV) trial for various types of acute respiratory failure in the emergency department; decreased mortality and use of the ICU. Respir Med. 2009 Jan;103(1):67-73. doi: 10.1016/j.rmed.2008.08.001. Epub 2008 Sep 18. PMID 18804357
- [Background] Chandra D, Stamm JA, Taylor B, Ramos RM, Satterwhite L, Krishnan JA, Mannino D, Sciurba FC, Holguin F. Outcomes of noninvasive ventilation for acute exacerbations of chronic obstructive pulmonary disease in the United States, 1998-2008. Am J Respir Crit Care Med. 2012 Jan 15;185(2):152-9. doi: 10.1164/rccm.201106-1094OC. Epub 2011 Oct 20. PMID 22016446
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Brochard L, Lefebvre JC, Cordioli RL, Akoumianaki E, Richard JC. Noninvasive ventilation for patients with hypoxemic acute respiratory failure. Semin Respir Crit Care Med. 2014 Aug;35(4):492-500. doi: 10.1055/s-0034-1383863. Epub 2014 Aug 11. PMID 25111645
- [Background] Rochwerg B, Brochard L, Elliott MW, Hess D, Hill NS, Nava S, Navalesi P Members Of The Steering Committee, Antonelli M, Brozek J, Conti G, Ferrer M, Guntupalli K, Jaber S, Keenan S, Mancebo J, Mehta S, Raoof S Members Of The Task Force. Official ERS/ATS clinical practice guidelines: noninvasive ventilation for acute respiratory failure. Eur Respir J. 2017 Aug 31;50(2):1602426. doi: 10.1183/13993003.02426-2016. Print 2017 Aug. PMID 28860265
- [Background] Vaschetto R, De Jong A, Conseil M, Galia F, Mahul M, Coisel Y, Prades A, Navalesi P, Jaber S. Comparative evaluation of three interfaces for non-invasive ventilation: a randomized cross-over design physiologic study on healthy volunteers. Crit Care. 2014 Jan 3;18(1):R2. doi: 10.1186/cc13175. PMID 24387642
- [Background] Navalesi P, Fanfulla F, Frigerio P, Gregoretti C, Nava S. Physiologic evaluation of noninvasive mechanical ventilation delivered with three types of masks in patients with chronic hypercapnic respiratory failure. Crit Care Med. 2000 Jun;28(6):1785-90. doi: 10.1097/00003246-200006000-00015. PMID 10890620
- [Background] Scala R, Accurso G, Ippolito M, Cortegiani A, Iozzo P, Vitale F, Guidelli L, Gregoretti C. Material and Technology: Back to the Future for the Choice of Interface for Non-Invasive Ventilation - A Concise Review. Respiration. 2020;99(9):800-817. doi: 10.1159/000509762. Epub 2020 Nov 18. PMID 33207357
- [Background] Crimi C, Noto A, Princi P, Esquinas A, Nava S. A European survey of noninvasive ventilation practices. Eur Respir J. 2010 Aug;36(2):362-9. doi: 10.1183/09031936.00123509. Epub 2010 Jan 14. PMID 20075052
- [Background] Lemyze M, Mallat J, Nigeon O, Barrailler S, Pepy F, Gasan G, Vangrunderbeeck N, Grosset P, Tronchon L, Thevenin D. Rescue therapy by switching to total face mask after failure of face mask-delivered noninvasive ventilation in do-not-intubate patients in acute respiratory failure. Crit Care Med. 2013 Feb;41(2):481-8. doi: 10.1097/CCM.0b013e31826ab4af. PMID 23263582
- [Background] Schallom M, Cracchiolo L, Falker A, Foster J, Hager J, Morehouse T, Watts P, Weems L, Kollef M. Pressure Ulcer Incidence in Patients Wearing Nasal-Oral Versus Full-Face Noninvasive Ventilation Masks. Am J Crit Care. 2015 Jul;24(4):349-56; quiz 357. doi: 10.4037/ajcc2015386. PMID 26134336
- [Background] Roberts CM, Brown JL, Reinhardt AK, Kaul S, Scales K, Mikelsons C, Reid K, Winter R, Young K, Restrick L, Plant PK. Non-invasive ventilation in chronic obstructive pulmonary disease: management of acute type 2 respiratory failure. Clin Med (Lond). 2008 Oct;8(5):517-21. doi: 10.7861/clinmedicine.8-5-517. PMID 18975486
- [Background] Antonelli M, Conti G, Pelosi P, Gregoretti C, Pennisi MA, Costa R, Severgnini P, Chiaranda M, Proietti R. New treatment of acute hypoxemic respiratory failure: noninvasive pressure support ventilation delivered by helmet--a pilot controlled trial. Crit Care Med. 2002 Mar;30(3):602-8. doi: 10.1097/00003246-200203000-00019. PMID 11990923
- [Background] Yamaguti WP, Moderno EV, Yamashita SY, Gomes TG, Maida AL, Kondo CS, de Salles IC, de Brito CM. Treatment-related risk factors for development of skin breakdown in subjects with acute respiratory failure undergoing noninvasive ventilation or CPAP. Respir Care. 2014 Oct;59(10):1530-6. doi: 10.4187/respcare.02942. Epub 2014 Jun 3. PMID 24894664
- [Background] Schettino G, Altobelli N, Kacmarek RM. Noninvasive positive pressure ventilation reverses acute respiratory failure in select "do-not-intubate" patients. Crit Care Med. 2005 Sep;33(9):1976-82. doi: 10.1097/01.ccm.0000178176.51024.82. PMID 16148468
- [Background] Conti G, Marino P, Cogliati A, Dell'Utri D, Lappa A, Rosa G, Gasparetto A. Noninvasive ventilation for the treatment of acute respiratory failure in patients with hematologic malignancies: a pilot study. Intensive Care Med. 1998 Dec;24(12):1283-8. doi: 10.1007/s001340050763. PMID 9885881
- [Background] Gorecki C, Brown JM, Nelson EA, Briggs M, Schoonhoven L, Dealey C, Defloor T, Nixon J; European Quality of Life Pressure Ulcer Project group. Impact of pressure ulcers on quality of life in older patients: a systematic review. J Am Geriatr Soc. 2009 Jul;57(7):1175-83. doi: 10.1111/j.1532-5415.2009.02307.x. Epub 2009 May 21. PMID 19486198
- [Background] Bennett G, Dealey C, Posnett J. The cost of pressure ulcers in the UK. Age Ageing. 2004 May;33(3):230-5. doi: 10.1093/ageing/afh086. PMID 15082426
- [Background] Drew P, Posnett J, Rusling L; Wound Care Audit Team. The cost of wound care for a local population in England. Int Wound J. 2007 Jun;4(2):149-55. doi: 10.1111/j.1742-481X.2007.00337.x. PMID 17651229
- [Background] Cai JY, Zha ML, Chen HL. Use of a Hydrocolloid Dressing in the Prevention of Device-related Pressure Ulcers During Noninvasive Ventilation: A Meta-analysis of Randomized Controlled Trials. Wound Manag Prev. 2019 Feb;65(2):30-38. PMID 30730303
- [Background] Davidson AC, Banham S, Elliott M, Kennedy D, Gelder C, Glossop A, Church AC, Creagh-Brown B, Dodd JW, Felton T, Foex B, Mansfield L, McDonnell L, Parker R, Patterson CM, Sovani M, Thomas L; BTS Standards of Care Committee Member, British Thoracic Society/Intensive Care Society Acute Hypercapnic Respiratory Failure Guideline Development Group, On behalf of the British Thoracic Society Standards of Care Committee. BTS/ICS guideline for the ventilatory management of acute hypercapnic respiratory failure in adults. Thorax. 2016 Apr;71 Suppl 2:ii1-35. doi: 10.1136/thoraxjnl-2015-208209. No abstract available. PMID 26976648
- [Background] Holanda MA, Reis RC, Winkeler GF, Fortaleza SC, Lima JW, Pereira ED. Influence of total face, facial and nasal masks on short-term adverse effects during noninvasive ventilation. J Bras Pneumol. 2009 Feb;35(2):164-73. doi: 10.1590/s1806-37132009000200010. PMID 19287920
- [Background] Cuvelier A, Pujol W, Pramil S, Molano LC, Viacroze C, Muir JF. Cephalic versus oronasal mask for noninvasive ventilation in acute hypercapnic respiratory failure. Intensive Care Med. 2009 Mar;35(3):519-26. doi: 10.1007/s00134-008-1327-x. Epub 2008 Oct 15. PMID 18854973
- [Background] Ozsancak A, Sidhom SS, Liesching TN, Howard W, Hill NS. Evaluation of the total face mask for noninvasive ventilation to treat acute respiratory failure. Chest. 2011 May;139(5):1034-1041. doi: 10.1378/chest.10-1905. Epub 2011 Feb 17. PMID 21330385
- [Background] Olivieri C, Costa R, Spinazzola G, Ferrone G, Longhini F, Cammarota G, Conti G, Navalesi P. Bench comparative evaluation of a new generation and standard helmet for delivering non-invasive ventilation. Intensive Care Med. 2013 Apr;39(4):734-8. doi: 10.1007/s00134-012-2765-z. Epub 2012 Dec 6. PMID 23223773
- [Background] Antonelli M, Pennisi MA, Pelosi P, Gregoretti C, Squadrone V, Rocco M, Cecchini L, Chiumello D, Severgnini P, Proietti R, Navalesi P, Conti G. Noninvasive positive pressure ventilation using a helmet in patients with acute exacerbation of chronic obstructive pulmonary disease: a feasibility study. Anesthesiology. 2004 Jan;100(1):16-24. doi: 10.1097/00000542-200401000-00007. PMID 14695719
- [Background] Antonaglia V, Ferluga M, Molino R, Lucangelo U, Peratoner A, Roman-Pognuz E, De Simoni L, Zin WA. Comparison of noninvasive ventilation by sequential use of mask and helmet versus mask in acute exacerbation of chronic obstructive pulmonary disease: a preliminary study. Respiration. 2011;82(2):148-54. doi: 10.1159/000324259. Epub 2011 Mar 26. PMID 21447934
- [Background] Longhini F, Liu L, Pan C, Xie J, Cammarota G, Bruni A, Garofalo E, Yang Y, Navalesi P, Qiu H. Neurally-Adjusted Ventilatory Assist for Noninvasive Ventilation via a Helmet in Subjects With COPD Exacerbation: A Physiologic Study. Respir Care. 2019 May;64(5):582-589. doi: 10.4187/respcare.06502. Epub 2019 Feb 12. PMID 30755472
- [Background] Pisani L, Mega C, Vaschetto R, Bellone A, Scala R, Cosentini R, Musti M, Del Forno M, Grassi M, Fasano L, Navalesi P, Nava S. Oronasal mask versus helmet in acute hypercapnic respiratory failure. Eur Respir J. 2015 Mar;45(3):691-9. doi: 10.1183/09031936.00053814. Epub 2014 Dec 10. PMID 25504992
- [Background] Girault C, Briel A, Benichou J, Hellot MF, Dachraoui F, Tamion F, Bonmarchand G. Interface strategy during noninvasive positive pressure ventilation for hypercapnic acute respiratory failure. Crit Care Med. 2009 Jan;37(1):124-31. doi: 10.1097/CCM.0b013e3181928706. PMID 19050635
- [Background] Vaschetto R, Turucz E, Dellapiazza F, Guido S, Colombo D, Cammarota G, Della Corte F, Antonelli M, Navalesi P. Noninvasive ventilation after early extubation in patients recovering from hypoxemic acute respiratory failure: a single-centre feasibility study. Intensive Care Med. 2012 Oct;38(10):1599-606. doi: 10.1007/s00134-012-2652-7. Epub 2012 Jul 24. PMID 22825283
- [Background] Newnam KM, McGrath JM, Salyer J, Estes T, Jallo N, Bass WT. A comparative effectiveness study of continuous positive airway pressure-related skin breakdown when using different nasal interfaces in the extremely low birth weight neonate. Appl Nurs Res. 2015 Feb;28(1):36-41. doi: 10.1016/j.apnr.2014.05.005. Epub 2014 Jun 5. PMID 25017108
- [Background] Bashir T, Murki S, Kiran S, Reddy VK, Oleti TP. 'Nasal mask' in comparison with 'nasal prongs' or 'rotation of nasal mask with nasal prongs' reduce the incidence of nasal injury in preterm neonates supported on nasal continuous positive airway pressure (nCPAP): A randomized controlled trial. PLoS One. 2019 Jan 31;14(1):e0211476. doi: 10.1371/journal.pone.0211476. eCollection 2019. PMID 30703172
- [Background] Vaschetto R, Longhini F, Persona P, Ori C, Stefani G, Liu S, Yi Y, Lu W, Yu T, Luo X, Tang R, Li M, Li J, Cammarota G, Bruni A, Garofalo E, Jin Z, Yan J, Zheng R, Yin J, Guido S, Della Corte F, Fontana T, Gregoretti C, Cortegiani A, Giarratano A, Montagnini C, Cavuto S, Qiu H, Navalesi P. Early extubation followed by immediate noninvasive ventilation vs. standard extubation in hypoxemic patients: a randomized clinical trial. Intensive Care Med. 2019 Jan;45(1):62-71. doi: 10.1007/s00134-018-5478-0. Epub 2018 Dec 10. PMID 30535516
- [Background] Curtis JR, Cook DJ, Sinuff T, White DB, Hill N, Keenan SP, Benditt JO, Kacmarek R, Kirchhoff KT, Levy MM; Society of Critical Care Medicine Palliative Noninvasive Positive VentilationTask Force. Noninvasive positive pressure ventilation in critical and palliative care settings: understanding the goals of therapy. Crit Care Med. 2007 Mar;35(3):932-9. doi: 10.1097/01.CCM.0000256725.73993.74. PMID 17255876
- [Background] da Cunha-Martins, B.S.M., Motta-Ribeiro, G.C. & Jandre, F.C. Short-term usage of three non-invasive ventilation interfaces causes progressive discomfort in healthy adults. Res. Biomed. Eng. 37, 289-298 (2021)
- [Background] Brill AK. How to avoid interface problems in acute noninvasive ventilation. Breathe 2014;10:230-242
- [Derived] Vaschetto R, Gregoretti C, Scotti L, De Vita N, Carlucci A, Cortegiani A, Crimi C, Mattei A, Scala R, Rocca E, Longhini F, Cammarota G, Misseri G, Dal Molin A, Scolletta S, Nava S, Maggiore SM, Navalesi P. A pragmatic, open-label, multi-center, randomized controlled clinical trial on the rotational use of interfaces vs standard of care in patients treated with noninvasive positive pressure ventilation for acute hypercapnic respiratory failure: the ROTAtional-USE of interface STUDY (ROTA-USE STUDY). Trials. 2023 Aug 13;24(1):527. doi: 10.1186/s13063-023-07560-1. PMID 37574558